CLINICAL TRIAL: NCT03393715
Title: Effect of Morning Versus Evening Perindopril on Blood Pressure Control in People With Type 2 Diabetes
Acronym: CHRONIC1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor of Endocrinology and Diabetes, Yaounde Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CNO20162
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Diabetes; Hypertension; Perindopril; chronobiology; Africa
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus | interventions — Perindopril

STUDY DESIGN:
Intervention Model Description: open label randomised controlled trial with crossover of perindopril administered in the morning versus evening on blood pressure control
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perindopril morning (Experimental): 10 mg of perindopril oral tablet once daily in the morning for 56 days
  Interventions: Drug: Perindopril Oral Tablet
- Perindopril evening (Active Comparator): 10 mg of perindopril oral tablet once daily in the evening for 56 days
  Interventions: Drug: Perindopril Oral Tablet

INTERVENTIONS:
Drug: Perindopril Oral Tablet — Perindopril oral tablet morning versus evening
  Other Names: Coversyl 10 mg

SUMMARY:
We assessed the influence of time of administration of ACE inhibitors on circadian blood pressure control in sub Saharan type 2 diabetes patients with stage 1 hypertension over 56 days as first line treatment.

DETAILED DESCRIPTION:
Background: Renin-angiotensin system antagonists represent the mainstay of blood pressure (BP) lowering treatment options in people with diabetes. ACE inhibitors have a long half-life and offer the advantage of a single daily dose, usually empirically taken in the morning.

Objective: We assessed the influence of time of administration of ACE inhibitors on circadian BP control in type 2 diabetes (T2D) patients with stage 1 hypertension.

Methods: Twenty T2D patients (9 being women) with a mean age of 58.7 years, diagnosed with stage 1 of hypertension and naive to BP lowering medications, were included. They were randomly allocated to receive perindopril 10 mg/day as a monotherapy either in the morning or in the evening for 28 days, with crossover without washout period on day 29th and additional 28 days follow-up. A 24-hour ambulatory BP monitoring (ABPM) was performed at baseline, days 28 and 56.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Grade 1 hypertension
* Informed consent

Exclusion Criteria:

* estimated creatinine clearance≤ 60ml/min
* White coat hypertension after initial 24 hour ABPM
* Previous antihypertensive treatment
* Pregnant women
* Individuals working during the night
* Hyperkalemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
24-hour blood pressure profile | 56 days
  Overall blood pressure control

SECONDARY OUTCOMES:
Night time blood pressure dip | 56 days
  Blood pressure drop at night

CONTACTS AND LOCATIONS:
Overall Officials: Eugène Sobngwi, MD, PhD, Principal Investigator — Yaounde Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided